CLINICAL TRIAL: NCT05451771
Title: An Open-label Phase I/II Trial of Venetoclax-Dexamethasone in Relapsed and/or Refractory t(11;14) Systemic Light-Chain Amyloidosis
Brief Title: Venetoclax-Dexamethasone in Relapsed and/or Refractory t(11;14) Amyloidosis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rajshekhar Chakraborty, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Rajshekhar Chakraborty, MD, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAT8639
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: AL Amyloidosis
Keywords: Light Chain Amyloidosis; Protein Misfolding Disorder
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Proteostasis Deficiencies | interventions — venetoclax; Dexamethasone; Calcium Dobesilate; daratumumab; Bendamustine Hydrochloride; pomalidomide; ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Phase 1: Venetoclax 200 mg (Experimental): Cohort 1: Venetoclax 200 mg tablet, once daily for up to 2 cycles after achieving best response, for a maximum of 6 cycles (1 cycle = 28 days)
  Interventions: Drug: Venetoclax Oral Tablet, 200 mg; Device: FISH assay
- Phase 1: Venetoclax 400mg (Experimental): Cohort 2: Venetoclax 400 mg tablet, once daily for up to 2 cycles after achieving best response, for a maximum of 6 cycles (1 cycle = 28 days)
  Interventions: Device: FISH assay; Drug: Venetoclax Oral Tablet, 400 mg
- Phase 1: Venetoclax 400mg + Dexamethasone 10 mg (Experimental): Cohort 3: Venetoclax 400 mg tablet, once daily and Dexamethasone 10 mg tablet once weekly, for up to 2 cycles after achieving best response, for a maximum of 6 cycles (1 cycle = 28 days)
  Interventions: Device: FISH assay; Drug: Venetoclax Oral Tablet, 400 mg; Drug: Dexamethasone Oral, 10 mg
- Phase 1: Venetoclax 400mg + Dexamethasone 20 mg (Experimental): Cohort 4: Venetoclax 400 mg tablet, once daily and Dexamethasone 20 mg tablet once weekly, for up to 2 cycles after achieving best response, for a maximum of 6 cycles (1 cycle = 28 days)
  Interventions: Device: FISH assay; Drug: Venetoclax Oral Tablet, 400 mg; Drug: Dexamethasone Oral, 20 mg
- Phase 2: Venetoclax MTD with Dexamethasone (Experimental): Venetoclax MTD (200 mg or 400 mg) with Dexamethasone (10 mg or 20 mg) as determined by the phase I results
  Interventions: Drug: Venetoclax MTD with Dexamethasone
- Phase 2: Control Arm (Investigator's Choice) (Active Comparator): Participants will receive one of the following as determined by the investigator:
  Daratumumab, Pomalidomide, Bendamustine, or Ixazomib (+/- dexamethasone)
  Interventions: Drug: Dexamethasone Oral, 20 mg; Drug: Daratumumab Injection; Drug: Bendamustine; Drug: Pomalidomide; Drug: Ixazomib

INTERVENTIONS:
Drug: Venetoclax Oral Tablet, 200 mg — 200 mg oral tablet daily
  Other Names: Venclexta
  Arms: Phase 1: Venetoclax 200 mg
Device: FISH assay — Cytogenetic analysis is intended for evaluation of relapsed/refractory AL amyloidosis using fluorescence in situ hybridization (FISH) using known translocation probes. Bone marrow aspirate (BMA) samples are collected in lavender top (Ethylenediaminetetraacetic acid (EDTA)) or green top (Sodium heparin) tubes. Specimen tubes shall be transported at room temperature to the laboratory on the same day of collection.
  Other Names: t(11;14) FISH assay
  Arms: Phase 1: Venetoclax 200 mg; Phase 1: Venetoclax 400mg; Phase 1: Venetoclax 400mg + Dexamethasone 10 mg; Phase 1: Venetoclax 400mg + Dexamethasone 20 mg
Drug: Venetoclax Oral Tablet, 400 mg — 400 mg oral tablet daily
  Other Names: Venclexta
  Arms: Phase 1: Venetoclax 400mg; Phase 1: Venetoclax 400mg + Dexamethasone 10 mg; Phase 1: Venetoclax 400mg + Dexamethasone 20 mg
Drug: Dexamethasone Oral, 10 mg — 10 mg oral tablet weekly
  Other Names: Decadron; Hemady
  Arms: Phase 1: Venetoclax 400mg + Dexamethasone 10 mg
Drug: Dexamethasone Oral, 20 mg — 20 mg oral tablet weekly
  Other Names: Decadron; Hemady
  Arms: Phase 1: Venetoclax 400mg + Dexamethasone 20 mg; Phase 2: Control Arm (Investigator's Choice)
Drug: Daratumumab Injection — Daratumumab will be administered at a dose of 16 mg/kg by IV infusion once weekly for weeks 1 to 8, every 2 weeks for weeks 9 to 24, and every 4 weeks thereafter for a maximum of 6 months of therapy. If subcutaneous formulation is available, participants can also receive subcutaneous daratumumab (1800 mg in 15 ml) in the same schedule.
  Other Names: Darzalex
  Arms: Phase 2: Control Arm (Investigator's Choice)
Drug: Bendamustine — Bendamustine will be given at an initial dose of 100 mg/m^2 intravenously on days 1 and 2 in each 28-day cycle.
  Other Names: Treanda
  Arms: Phase 2: Control Arm (Investigator's Choice)
Drug: Pomalidomide — Pomalidomide will be administered at an initial dose of 2 mg per days on days 1-21 every 28 days.
  Other Names: Pomalyst
  Arms: Phase 2: Control Arm (Investigator's Choice)
Drug: Ixazomib — Ixazomib will be administered at an initial dose of 4 mg per days on days 1, 8, and 15 every 28 days.
  Other Names: Ninlaro
  Arms: Phase 2: Control Arm (Investigator's Choice)
Drug: Venetoclax MTD with Dexamethasone — Venetoclax MTD (200 mg or 400 mg) with Dexamethasone (10 mg or 20 mg) as determined by the phase I results
  Arms: Phase 2: Venetoclax MTD with Dexamethasone

SUMMARY:
The purpose of this study is assess safety, safest dose, and effectiveness of venetoclax in combination with dexamethasone in participants with t(11;14) positive relapsed (comes back) or refractory (did not get better) light chain amyloidosis.

DETAILED DESCRIPTION:
This study is a phase 1/2 study of venetoclax-dexamethasone combination therapy in relapsed/refractory t(11;14) systemic immunoglobulin light chain amyloidosis (AL) amyloidosis. The phase 1 is a dose escalation designed to determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of venetoclax in combination with low-dose weekly dexamethasone. There will be four candidate-dosing cohorts of venetoclax with or without dexamethasone in the Phase I dose-escalation. Dose escalation will be guided by the Bayesian optimal interval (BOIN) design with accelerated titration up to a total sample size of 15 participants.

The phase 2 portion is a randomized open-label study comparing the MTD or RP2D of venetoclax in combination with dexamethasone versus investigator's choice (daratumumab, pomalidomide, bendamustine, or ixazomib (with or without dexamethasone).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of signing Informed Consent Form
* Ability to comply with the study protocol, in the investigator's judgment
* Confirmed diagnosis of systemic AL amyloidosis by mass spectrometry or immunohistochemistry (IHC) on a tissue biopsy
* Has received ≥1 prior lines of therapy, including an anti-cluster of differentiation 38 (CD 38) monoclonal antibody
* Participants with a history of autologous hematopoietic cell transplantation must have recovered from any transplant-related toxicities
* Presence of t(11;14) on FISH at any time since diagnosis (Eligibility must confirmed by FISH testing at Columbia University Irving Medical Center (CUIMC)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2

Exclusion Criteria:

* Known hypersensitivity to any of the study drugs
* History of other malignancy that could affect compliance with the protocol or interpretation of results (Patients with a history of curatively treated basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix, breast cancer, or Hodgkin's Lymphoma are generally eligible. Patients with a malignancy that has been treated, but not with curative intent, will be excluded, unless the malignancy has been in remission without treatment for ≥ 2 years prior to enrollment.)
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to, uncontrolled systemic infection (viral, bacterial, or fungal)
* Patients on renal replacement therapy
* Known GI disease or GI procedure that could interfere with oral absorption (including difficulty swallowing)
* New York Heart Association (NYHA) Class III or IV heart failure
* Mayo stage three-B (IIIB) with N-terminal pro-hormone B-type natriuretic peptide (NT-Pro BNP) > 8500 pg/mL
* Prior exposure to anti-apoptotic protein B-cell lymphoma 2 (BCL-2) inhibitors
* Patients with human immunodeficiency virus (HIV) who are not on highly active antiretroviral therapy (HAART) or those with active hepatitis A, B, or C infection
* Patients meeting criteria for symptomatic multiple myeloma by one of the following:(a) Lytic lesions on imaging (b) Plasmacytoma, (c) Hypercalcemia without any alternate etiology, or (c) Bone marrow plasma cell infiltrate of greater than 60%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLT) (Phase 1) | Up to 6 cycles (approximately 6 months)
  The number of participants with dose limiting toxicities for each treatment dose will be used to determine the MTD. Dose limiting toxicity defined as grade 4 neutropenia lasting more than 5 days, any grade febrile neutropenia, grade 4 thrombocytopenia, grade 3 thrombocytopenia with bleeding, other therapy related non-hematologic toxicity of grade 2 or higher that requires discontinuation of therapy, clinical tumor lysis syndrome (TLS), laboratory TLS if the metabolic abnormalities are considered clinically significant by the investigator. All other grade 3 or higher adverse events (AEs) will be considered as DLTs with a few exceptions.
Hematologic ≥ Very Good Partial Response (VGPR) Rate (Phase 2) | Up to 6 cycles (approximately 6 months)
  Hematologic ≥VGPR rate defined as proportion of participants achieving VGPR, low serum differential free light chain concentration (dFLC) partial response (PR), or a complete (CR).
  VGPR is defined as the difference between involved and uninvolved free light chain (FLC) [dFLC] < 40 mg/L. Low dFLC PR is defined as achieving a dFLC<10 mg/L, low dFLC PR will be considered as a deep hematologic response and included in the ≥VGPR category). CR is defined as negative serum and urine immunofixation electrophoresis along with a serum free light chain ratio that lies within the normal range or skewed towards the non-amyloid forming light chain, as per institutional laboratory values

SECONDARY OUTCOMES:
Overall Organ Response Rate (ORR) (Phase 2) | Up to 1 year
  ORR defined as proportion of evaluable participants achieving organ response in each involved organ
Progression Free Survival (PFS) (Phase 2) | Up to 1 year
  PFS defined as time from the date of enrollment to hematologic progression or death, whichever is earlier
Overall Hematologic Response Rate (HRR) (Phase 2) | Up to 1 year
  HRR defined as proportion of patients achieving partial response (PR) or better
Duration of Hematologic Response (DOHR) (Phase 2) | Up to 1 year
  DOHR defined as time from the date of first documentation of hematologic response to the date of first documented hematologic disease progression
Time to hematologic ≥VGPR (Phase 2) | Up to 1 year
  Time to hematologic ≥VGPR defined as time from the first dose of study treatment to achievement of deep hematologic response (VGPR, low dFLC PR, or a CR)
Time to next treatment (TTNT) (Phase 2) | Up to 1 year
  TTNT defined as time from the date of enrollment to initiation of a subsequent line of therapy
Major Organ Deterioration-Progression Free Survival (MOD-PFS) (Phase 2) | Up to 1 year
  MOD-PFS defined as time from the date of enrollment to one of the following events (whichever occurs first): death, clinical manifestation of cardiac/renal failure, or development of hematologic progression of disease
Overall Survival (OS) (Phase 2) | Up to 1 year
  OS defined as the time from the date of enrollment to death from any cause
Patient-reported outcomes (PROs) (Phase 2) | Start of each cycle (Day 1 of each 28 day cycle) and Follow-up (every 8 weeks for up to 1 year)
  PROs defined as longitudinal score of "Physical Functioning" domain of Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Profile v2.0 The Physical Functioning domain contains four items with a 1 (unable to do) to 5 (without any difficulty) numeric rating.

CONTACTS AND LOCATIONS:
Overall Officials: Rajshekhar Chakraborty, MD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - Boston Medical Center, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - New York Presbyterian Hospital/Columbia University Irving Medical Center, New York, New York
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Locke M, Nieto M. AL Amyloidosis: Current Treatment and Outcomes. Adv Hematol. 2025 Mar 3;2025:7280805. doi: 10.1155/ah/7280805. eCollection 2025. PMID 40226119